CLINICAL TRIAL: NCT00162487
Title: Evaluation of β2 Genetic Polymorphisms and the Effect of Albuterol Inhalation on Potassium and Glucose Plasma Concentration
Brief Title: Genetic Determinants of the Hypokalemic and Hyperglycemic Effect of Albuterol Inhalation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yc19556-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Hyperkalemia; Chronic Renal Failure
MeSH Terms: conditions — Hyperkalemia; Kidney Failure, Chronic | interventions — Albuterol

INTERVENTIONS:
Drug: Albuterol (1,200 μg) through metered-dose inhaler

SUMMARY:
Several studies have indicated that albuterol administered either intravenously or by inhalation can significantly reduce plasma potassium concentration in patients suffering from chronic renal failure.In conjunction with the decrease in potassium concentration a modest rise in glucose concentration is usually noted. These metabolic effects are characterized by rapid onset occurring as early as 3-5 minutes following salbutamol administration and lasting for at least 1 hour.

The role played by ß2AR polymorphisms in determining the bronchial and vascular response to ß2AR agonist drugs, have been confirmed by several studies.

The purpose of the present study is to examine possible causal relationships between genetically based alteration in the structure of ß2AR and the metabolic effects of inhaled albuterol.

ELIGIBILITY:
Inclusion Criteria:

* patients regularly attending the nephrological clinic or the dialysis unit
* persistent potassium concentration above 5 mEq/L

Exclusion Criteria:

1. Patients suffering from active ischemic heart disease
2. Patient with a recent history of arrhythmia
3. Patients treated regularly with ß blockers
4. Patients treated regularly with salbutamol or other ß2AR agonists
5. Patients suffering from persistent tachycardia (pulse > 100 beats/min)
6. Patients who are hemodynamically unstable
7. Patients suffering from any acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-08

PRIMARY OUTCOMES:
The extent of decrease in plasma potassium concentration
The extent of increase in plasma glucose concentration
Plasma concentration of albuterol

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel